CLINICAL TRIAL: NCT06471309
Title: Effect of Theta Burst Transcranial Magnetic Stimulation on Post-Stroke Dysphagia
Brief Title: Effect of Theta Burst Transcranial Magnetic Stimulation on Patients with Dysphagia After Stroke
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Xiaohui (Other)
Responsible Party: Sponsor-Investigator, Zhang Xiaohui, sponsor, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240619
Record Dates: First submitted 2024-06-19; First posted 2024-06-24 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Dysphagia; Functional Near- Infrared Spectroscopy; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bilateral stimulation group (Experimental): On the basis of routine treatment and routine swallowing rehabilitation training, iTBS treatment was given to the representative area of mylohyoid cortex on the affected side and cTBS treatment was given to the representative area of mylohyoid cortex on the healthy side
  Interventions: Device: Theta burst transcranial magnetic stimulation
- Unilateral stimulation group (Experimental): On the basis of routine treatment and routine swallowing rehabilitation training, iTBS treatment was given to the representative area of mylohyoid cortex on the affected side and sham cTBS treatment was given to the representative area of mylohyoid cortex on the healthy side
  Interventions: Device: Theta burst transcranial magnetic stimulation
- Sham stimulation group (Sham Comparator): On the basis of routine treatment and routine swallowing rehabilitation training, sham iTBS treatment was given to the representative area of mylohyoid cortex on the affected side and sham cTBS treatment was given to the representative area of mylohyoid cortex on the healthy side
  Interventions: Device: Theta burst transcranial magnetic stimulation

INTERVENTIONS:
Device: Theta burst transcranial magnetic stimulation — The stimulation intensity of TBS was 80%RMT, with a total of 600 pulses, five times a week for two weeks. In the bilateral stimulation group, iTBS treatment was given to the representative area of mylohyoid cortex on the affected side and cTBS treatment was given to the representative area of mylohyoid cortex on the healthy side. In the unilateral stimulation group, iTBS treatment was given to the representative area of mylohyoid cortex on the affected side and sham cTBS treatment was given to the representative area of mylohyoid cortex on the healthy side. In the sham stimulation group, sham iTBS treatment was given to the representative area of mylohyoid cortex on the affected side and sham cTBS treatment was given to the representative area of mylohyoid cortex on the healthy side. When giving sham stimulation, put the coil vertically so that the coil is perpendicular to the patient's skull surface , it will not produce real therapeutic effect.

SUMMARY:
The purpose of this study was to observe the effect of Theta burst transcranial magnetic stimulation (TBS) on swallowing function in patients with dysphagia after stroke (PSD). Functional near- infrared spectroscopy (fNIRS) was used to detect the changes in activation and functional connectivity of related brain regions in PSD patients treated with intermittent TBS（iTBS）stimulation on the affected side and consistent TBS（cTBS） stimulation on the healthy side. To investigate the effects of TBS on swallowing related cortical excitability in stroke patients with dysphagia and explore its possible mechanism, and provide theoretical basis for the treatment of PSD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* The first stroke lasted from 2 weeks to 6 months, with stable vital signs and right-handedness
* The stroke met the diagnostic criteria of "Chinese Guidelines for the Diagnosis and Treatment of Cerebral Hemorrhage 2019" or "Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018" formulated by the Cerebrovascular Department of the Branch of Neurology of the Chinese Medical Association, and the cerebral CT or MRI examination showed unilateral cerebral infarction or cerebral hemorrhage.
* The dysphagia was consistent with the Expert Consensus on the Evaluation and Treatment of dysphagia in China (2017 edition), and the dysphagia was confirmed by videofluoroscopic swallowing study.
* MMSE>24, good cognitive function
* The skull is intact without craniotomy or repair
* Subject or family members sign informed consent

Exclusion Criteria:

* Combined with other diseases that may cause swallowing disorders, such as Parkinson's disease, dementia, motor neurone disease and other neurological diseases, or esophageal, neck surgery and other diseases that cause swallowing organ structure abnormalities
* A history of mental illness or epilepsy
* A metal implant in the head or eye, a pacemaker or a drug pump in the body
* Pregnancy, malignant tumor, serious disease history of heart, liver, kidney and other important organs
* Ulceration or infection of the skin on the head or where the electrode is applied
* Poor compliance and inability to complete basic treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Rosenbek Penetration-aspiration scale | The first evaluation was before the intervention and the second evaluation was after 2 weeks of treatment.
  The Rosenbek Penetration-aspiration scale assesses the patient's swallowing function by assessing the severity of penetration and aspiration. The results of Rosenbek Penetration-aspiration scale are divided into 8 grades from 1 to 8, and the lower the score, the better the swallowing ability.
Standardized Swallowing Assessment | The first evaluation was before the intervention and the second evaluation was after 2 weeks of treatment.
  The Standardized Swallowing Assessment scale is divided into three parts: clinical examination, water test, and normal eating, and is used to evaluate the safety and effectiveness of swallowing. The highest score of Standardized Swallowing Assessment scale is 46, and the lowest score is 18. The lower the score, the better the swallowing function.
functional near- infrared spectroscopy | The first evaluation was before the intervention and the second evaluation was after 2 weeks of treatment.
  fNIRS is a brain function detection technology, which can indirectly reflect the brain neural activity by detecting the content of oxygenated and deoxygenated hemoglobin in the cerebral cortex in real time. In this study, fNIRS was used to assess brain region activation and network connectivity characteristics during swallowing tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No